CLINICAL TRIAL: NCT03925220
Title: Testing a Brief Substance Misuse Preventative Intervention for Parents of Youth
Brief Title: Testing a Brief Substance Misuse Preventative Intervention for Parents/Guardians of 5th-7th Grade Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Margie Skeer, Associate Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01DA045073-01A1 (NIH)
Record Dates: First submitted 2019-04-08; First posted 2019-04-24 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Substance-Related Disorders; Underage Drinking; Drug Use
Keywords: Primary Prevention; Adolescent Behavior; Family; Personal Communication
MeSH Terms: conditions — Substance-Related Disorders; Underage Drinking; Adolescent Behavior; Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Substance Use Prevention Intervention (Experimental): Parents will be given a handbook specific to the gender of their child that provides information and advice communication and substance use prevention. Parents will then participate in a one-hour session with an interventionist where the main points in the handbook will be reviewed and they will fill out an action plan on how to make changes in communication about substances with their child. The interventionist will also provide parents with a referral packet. Two weeks after the live session, participants will have a half-hour follow-up phone call with the same study interventionist. For the home-based component, parents will receive two messages each week with reminders and tips that reinforce the information covered in the handbook. Finally, participants will receive a magnet about the importance of family meals that they will be instructed to put on their refrigerators.
  Interventions: Behavioral: The SUPPER Project
- Nutrition, Physical Activity, and Weight Talk Comparison (Active Comparator): For the comparison condition, after the baseline assessment, parents will receive a handbook on nutrition and physical activity entitled: "Healthy Eating & Physical Activity Across Your Lifespan: Helping your Child - Tips for Parents". This handbook, which is adapted from the handbook developed by the National Institute of Diabetes and Digestive and Kidney Diseases and the Weight Control Information Network, is approximately the same length as the intervention handbook and is available in English and Spanish. It is given with an insert on reducing weight talk and weight teasing in the family. Parents will also receive a magnet with a message about nutrition and exercise. To control for contact time, these participants will meet live with a study staff member two weeks after receiving the handbook, complete an action plan, and have the 30-minute call, as well as receive two text messages twice per week for 13 weeks with tips and reminders from the comparison handbook and insert.
  Interventions: Behavioral: Improving nutrition and physical activity among youth

INTERVENTIONS:
Behavioral: The SUPPER Project — Substance Use Promoted by Eating family meals Regularly
  Arms: Substance Use Prevention Intervention
Behavioral: Improving nutrition and physical activity among youth — A brief intervention focused on improving nutrition and physical activity among youth
  Arms: Nutrition, Physical Activity, and Weight Talk Comparison

SUMMARY:
The current study aims to test the efficacy of a family communication-based, novel, adaptable, and resource-efficient substance misuse preventive intervention for parents/guardians of pre/early adolescents (grades 5-7). The short-term goal of this study is to increase the quality time that parents spend with their children through eating meals together, and in so doing, talking about the harms associated with substance use (intermediate endpoint), which will in turn, lead to the long-term goal of preventing the initiation and misuse of substances among their children as they enter adolescence.

DETAILED DESCRIPTION:
The prevention of substance use and misuse among adolescents is a national public health priority. Universal prevention programs that include parents/guardians (referred to as "parents") in this effort have been shown to prevent and reduce substance use problems among adolescents. However, the programs that have been most effective are resource and participant intensive. In addition, the majority of the current programs are not gender-specific and in some cases, long-term effects have been shown for one gender but not the other. The purpose of the current study is to test the efficacy of a brief, communication-based, substance use preventive intervention for parents of pre/early adolescents. The proposal is based on data from a study funded by the National Institute on Drug Abuse (NIDA) where the investigative team conducted a pilot randomized controlled trial (RCT) of the intervention among 70 parents/guardians and their children. The intervention was found to be acceptable and feasible to participants and families in the intervention had increased parent-child communication about substance use compared to those in the control condition. The purpose of the pilot study was to lay the groundwork for a large-scale trial of the intervention with 500 parent-child dyads. The brief intervention framework utilizes a one-time live (in person or remote) session and a follow-up phone call with a communication specialist to facilitate parents' roles as preventionists, which will focus on family interactions at meals, the role of peers in substance use, and parent-child communication about substance use. For this live session, parents will be asked to review a handbook with gender-specific information that emphasizes engaging in family meals, communication, and talking with their child about the harms of substance use. For the home-based component, tips and reminders with content from the handbooks will be sent via text messages throughout the three-month study period. Parents in the comparison condition will receive a handbook, similar in length and structure, on nutrition and physical activity, as well as receive comparison text messages and meet with a study team member. All study materials will be available in English and Spanish. It is hypothesized that over the study period, parents randomized to the intervention will have an increased frequency of parent-child communication about substance use. It is also hypothesized that these parents will have more positive and fewer negative family interactions during meals and qualitatively better content of conversations about substance use with their children compared to parents in the comparison condition. Furthermore, it is hypothesized that compared to children of parents in the comparison condition, children of parents who receive the intervention will self-report reduced intentions and willingness to use substances, reduced affiliation with substance-using peers, and increased negative attitudes and expectancies regarding substance use, and secondarily, lower rates of substance use initiation.

ELIGIBILITY:
Inclusion Criteria:

* The parent/guardian must have a child between 5th-7th grades at the start of the project;
* The parent must be the custodial parent, living with the child at least 50% of the time (as in the case of joint custody); and
* Parental consent and child assent are obtained.

Exclusion Criteria:

* Parents of children with self-identified developmental disabilities who would have difficulty understanding the baseline assessment; and
* Parents or families who are not able to speak, read, and understand English or Spanish well enough to complete study procedures.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 402 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margie Skeer, ScD, MPH, MSW, Principal Investigator — Tufts University School of Medicine
Locations (1):
- Tufts University School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Skeer MR, Sabelli RA, Rancano KM, Lee-Bravatti M, Ryan EC, Eliasziw M, Spirito A. Randomized controlled trial to test the efficacy of a brief, communication-based, substance use preventive intervention for parents of adolescents: Protocol for the SUPPER Project (Substance Use Prevention Promoted by Eating family meals Regularly). PLoS One. 2022 Feb 2;17(2):e0263016. doi: 10.1371/journal.pone.0263016. eCollection 2022. PMID 35108294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol enrollment reflects the number of parent and child dyads enrolled in the study. Before COVID-19, participants were recruited through schools. After COVID-19, participants were recruited through community-based organizations and an online recruitment company.
Pre-assignment Details: Participants were screened for eligibility and had to complete all baseline assessments. Parents and children were eligible to participate if: (1) the child was enrolled in 5th, 6th, or 7th grade at a school within Massachusetts at the time of recruitment, (2) the child and parent were able to independently complete study activities in English or Spanish, (3) the parent and child were living together at least 50% of the time, (4) parents consent to participate and child gives assent.
Groups:
- Substance Use Prevention Intervention - Parents: Parents were given a handbook specific to the gender of their child that provides information and advice on communication and substance use prevention. Parents then participated in a one-hour session with an interventionist where the main points in the handbook were reviewed and they filled out an action plan on how to make changes in communication about substances with their child. The interventionist also provided parents with a referral packet. Two weeks after the live session, participants had a half-hour follow-up phone call with the same study interventionist. For the home-based component, parents received two messages each week with reminders and tips that reinforce the information covered in the handbook. Finally, participants received a magnet about the importance of family meals that they were instructed to put on their refrigerators.
- Substance Use Prevention Intervention - Children: Children discussed with their parents a handbook specific to their gender that provides information and advice on communication and substance use prevention. Children participated with their parents in completing an action plan on how to make changes in communication about substances. Children received reminders and tips that reinforce the information covered in the handbook. Finally, participants received a magnet about the importance of family meals that they were instructed to put on their refrigerators.
- Nutrition, Physical Activity, and Weight Talk Comparison - Parents: Parents received a handbook on nutrition and physical activity entitled: "Healthy Eating & Physical Activity Across Your Lifespan: Helping your Child - Tips for Parents". This handbook, which is adapted from the handbook developed by the National Institute of Diabetes and Digestive and Kidney Diseases and the Weight Control Information Network, is approximately the same length as the intervention handbook and is available in English and Spanish. It is given with an insert on reducing weight talk and weight teasing in the family. Parents also received a magnet with a message about nutrition and exercise. To control for contact time, these participants met live with a study staff member two weeks after receiving the handbook, completed an action plan, and had the 30-minute call, as well as receive two text messages twice per week for 13 weeks with tips and reminders from the comparison handbook and insert.
- Nutrition, Physical Activity, and Weight Talk Comparison - Children: Children discussed with their parents a handbook on nutrition and physical activity entitled: "Healthy Eating & Physical Activity Across Your Lifespan: Helping your Child - Tips for Parents". This handbook, which is adapted from the handbook developed by the National Institute of Diabetes and Digestive and Kidney Diseases and the Weight Control Information Network, is approximately the same length as the intervention handbook and is available in English and Spanish. It is given with an insert on reducing weight talk and weight teasing in the family. Participants also received a magnet with a message about nutrition and exercise. Children also helped their parents complete an action plan and received tips and reminders from the comparison handbook and insert.
Period: Overall Study
Arm/Group | Substance Use Prevention Intervention - Parents | Substance Use Prevention Intervention - Children | Nutrition, Physical Activity, and Weight Talk Comparison - Parents | Nutrition, Physical Activity, and Weight Talk Comparison - Children
Started (The number of participants enrolled (completed informed consent and assent, and completed baseline submissions) and randomized.) | 201 | 201 | 201 | 201
Baseline Analyzed (The number of participants who completed baseline and one or more follow-up surveys.) | 192 | 192 | 196 | 196
3 Months Follow-up | 181 | 181 | 185 | 185
6 Months Follow-up | 159 | 159 | 170 | 170
12 Months Follow-up | 152 | 148 | 150 | 150
18 Months Follow-up | 157 | 151 | 160 | 159
Completed | 157 | 151 | 160 | 159
Not Completed | 44 | 50 | 41 | 42
Not completed — Withdrawal by Subject | 4 | 4 | 4 | 4
Not completed — Lost to Follow-up | 40 | 46 | 37 | 38

BASELINE CHARACTERISTICS:
Population: The overall number of participants at baseline includes parent and child participants who completed one or more post-randomization surveys.
Groups:
- Substance Use Prevention Intervention: Parents were given a handbook specific to the gender of their child that provides information and advice communication and substance use prevention. Parents then participated in a one-hour session with an interventionist where the main points in the handbook were reviewed and they filled out an action plan on how to make changes in communication about substances with their child. The interventionist also provided parents with a referral packet. Two weeks after the live session, participants had a half-hour follow-up phone call with the same study interventionist. For the home-based component, parents received two messages each week with reminders and tips that reinforce the information covered in the handbook. Finally, participants received a magnet about the importance of family meals that they were instructed to put on their refrigerators.
- Nutrition, Physical Activity, and Weight Talk Comparison: For the comparison condition, after the baseline assessment, parents received a handbook on nutrition and physical activity entitled: "Healthy Eating & Physical Activity Across Your Lifespan: Helping your Child - Tips for Parents". This handbook, which is adapted from the handbook developed by the National Institute of Diabetes and Digestive and Kidney Diseases and the Weight Control Information Network, is approximately the same length as the intervention handbook and is available in English and Spanish. It is given with an insert on reducing weight talk and weight teasing in the family. Parents also received a magnet with a message about nutrition and exercise. To control for contact time, these participants met live with a study staff member two weeks after receiving the handbook, completed an action plan, and had the 30-minute call, as well as receive two text messages twice per week for 13 weeks with tips and reminders from the comparison handbook and insert.
- Total: Total of all reporting groups
Arm/Group | Substance Use Prevention Intervention | Substance Use Prevention Intervention - Children | Nutrition, Physical Activity, and Weight Talk Comparison | Nutrition, Physical Activity, and Weight Talk Comparison - Children | Total
Number analyzed (Participants) | 192 | 192 | 196 | 196 | 776
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was calculated by date of birth and date of survey completion.
  years | 42.1 (6.3) | 11.8 (1.1) | 43.3 (6.8) | 11.8 (1.0) | 27.3 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex was measured by asking about biological sex assigned at birth.
  Participants
    Female | 169 | 99 | 173 | 102 | 543
    Male | 23 | 93 | 23 | 94 | 233
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was measured by asking "Do you consider yourself Hispanic or Latino/a?".
  Participants
    Hispanic or Latino | 41 | 48 | 40 | 42 | 171
    Not Hispanic or Latino | 151 | 144 | 156 | 154 | 605
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was measured by asking "Which of the following best describes you?".
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 8 | 9 | 7 | 4 | 28
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 1 | 3
    Black or African American | 19 | 21 | 26 | 28 | 94
    White | 117 | 104 | 118 | 110 | 449
    More than one race | 7 | 9 | 4 | 11 | 31
    Unknown or Not Reported | 41 | 48 | 40 | 42 | 171
Region of Enrollment [Count of Participants; unit: Participants] — Participants were asked in which school district the child attends school.
  Participants
    United States | 192 | 192 | 196 | 196 | 776
Frequency of parent-child conversations on substances [Count of Participants; unit: Participants] — Frequency of conversations was measured using an item adapted from a measure for parent-child communication about sex (Miller et al, 1998).
  Question: "During the past 3-months, how many times have you and your child talked about [substance]?" The same question assessed frequency for each substance of interest (alcohol, cigarettes, e-cigarettes, cannabis, other drugs) on a five-point Likert scale from "None" to "A lot". Responses were dichotomized as "Several" or "A lot" versus "None", "Once", or "A few times". Population: Missing participants did not answer the survey question.
  Participants
    On drinking alcohol: 'Several times' or 'a lot' | 28 | 17 | 36 | 23 | 104
    On drinking alcohol: 'None', 'once', or 'a few times' | 164 | 175 | 160 | 173 | 672
    On smoking cigarettes: 'Several times' or 'a lot' | 23 | 12 | 26 | 19 | 80
    On smoking cigarettes: 'None', 'once', or 'a few times' | 169 | 180 | 170 | 177 | 696
    On using cannabis: 'Several times' or 'a lot' | 16 | 14 | 27 | 18 | 75
    On using cannabis: 'None', 'once', or 'a few times' | 176 | 178 | 169 | 178 | 701
    On vaping: 'Several times' or 'a lot' | 19 | 14 | 31 | 13 | 77
    On vaping: 'None', 'once', or 'a few times' | 173 | 178 | 165 | 183 | 699
    On using other drugs: 'Several times' or 'a lot' | 23 | 17 | 23 | 25 | 88
    On using other drugs: 'None', 'once', or 'a few times' | 169 | 175 | 173 | 171 | 688
Targeted parent-child communication on substance use [Count of Participants; unit: Participants] — An adapted version of the Targeted Parent-Child Communication about Alcohol Scale (Miller-Day et al, 2010) was used to assess targeted communication about alcohol and other drugs use. The ten-item assesses parents' agreement on having communication about substance use related topics and applying strategies parents may have discussed with their child. Items were assessed on a six-point Likert scale from "Strongly agree" to "Strongly disagree". Responses were dichotomized as "Agree" or "Strongly Agree" versus "Strongly Disagree" to "Somewhat Agree".
  Participants
    Warned about the dangers: Agree | 142 | 164 | 157 | 168 | 631
    Warned about the dangers: Disagree | 50 | 28 | 39 | 28 | 145
    Talked about how to handle offers: Agree | 81 | 122 | 88 | 116 | 407
    Talked about how to handle offers: Disagree | 111 | 70 | 108 | 80 | 369
    Given rules to obey: Agree | 72 | 115 | 82 | 111 | 380
    Given rules to obey: Disagree | 120 | 77 | 114 | 85 | 396
    Not directly talked but given hints: Agree | 44 | 58 | 41 | 64 | 207
    Not directly talked but given hints: Disagree | 148 | 134 | 155 | 132 | 569
    Lectured or given speech: Agree | 69 | 84 | 66 | 88 | 307
    Lectured or given speech: Disagree | 123 | 108 | 130 | 108 | 469
    Made a comment on character on TV: Agree | 69 | 70 | 78 | 73 | 290
    Made a comment on character on TV: Disagree | 123 | 122 | 118 | 123 | 486
    Told stories of people: Agree | 104 | 58 | 104 | 75 | 341
    Told stories of people: Disagree | 88 | 134 | 92 | 121 | 435
    Told they would be disappointed: Agree | 49 | 91 | 57 | 95 | 292
    Told they would be disappointed: Disagree | 143 | 101 | 139 | 101 | 484
    Shown information about the dangers: Agree | 53 | 50 | 47 | 59 | 209
    Shown information about the dangers: Disagree | 139 | 142 | 149 | 137 | 567
    Asked about their thoughts/opinions: Agree | 102 | 106 | 107 | 115 | 430
    Asked about their thoughts/opinions: Disagree | 90 | 86 | 89 | 81 | 346

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Parent-child Conversations on Substances
Description: Frequency of conversations was measured using an item adapted from a measure for parent-child communication about sex (Miller et al, 1998).
  Question: "During the past 3-months, how many times have you and your child talked about [substance]?" The same question assessed frequency for each substance of interest (alcohol, cigarettes, e-cigarettes, cannabis, other drugs) on a five-point Likert scale from "None" to "A lot". Responses were dichotomized as "Several" or "A lot" versus "None", "Once", or "A few times".
  This measure was reported by parents and children.
Time Frame: 3 months (short-term) and 18 months (long-term)
Population: Sample sizes differ for parent- and child-reported data based on how many parents and children completed the survey at each follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Substance Use Prevention Intervention | Substance Use Prevention Intervention - Children | Nutrition, Physical Activity, and Weight Talk Comparison | Nutrition, Physical Activity, and Weight Talk Comparison - Children
Number analyzed (Participants) | 178 | 178 | 185 | 185
Participants
  3-months - drinking alcohol: 'Several times' or 'a lot' | 87 | 32 | 29 | 20
  3-months - drinking alcohol: 'None', 'once', or 'a few times' | 91 | 146 | 156 | 165
  3-months - using e-cigarettes or vaping: 'Several times' or 'a lot' | 70 | 28 | 28 | 17
  3-months - using e-cigarettes or vaping: 'None', 'once', or 'a few times' | 108 | 150 | 157 | 168
  3-months - using marijuana: 'Several times' or 'a lot' | 61 | 20 | 27 | 17
  3-months - using marijuana: 'None', 'once', or 'a few times' | 117 | 158 | 158 | 168
  3-months - smoking cigarettes: 'Several times' or 'a lot' | 79 | 28 | 23 | 21
  3-months - smoking cigarettes: 'None', 'once', or 'a few times' | 99 | 150 | 162 | 164
  3-months - using other drugs: 'Several times' or 'a lot' | 55 | 25 | 20 | 19
  3-months - using other drugs: 'None', 'once', or 'a few times' | 123 | 153 | 165 | 166
  18-months - drinking alcohol: number analyzed (Participants) | 157 | 151 | 160 | 159
  18-months - drinking alcohol: 'Several times' or 'a lot' | 51 | 30 | 36 | 28
  18-months - drinking alcohol: 'None', 'once', or 'a few times' | 106 | 121 | 124 | 131
  18-months - using e-cigarettes or vaping: number analyzed (Participants) | 157 | 151 | 160 | 159
  18-months - using e-cigarettes or vaping: 'Several times' or 'a lot' | 40 | 22 | 33 | 18
  18-months - using e-cigarettes or vaping: 'None', 'once', or 'a few times' | 117 | 129 | 127 | 141
  18-months - using marijuana: number analyzed (Participants) | 157 | 151 | 160 | 159
  18-months - using marijuana: 'Several times' or 'a lot' | 38 | 26 | 30 | 22
  18-months - using marijuana: 'None', 'once', or 'a few times' | 119 | 125 | 130 | 137
  18-months - smoking cigarettes: number analyzed (Participants) | 157 | 151 | 160 | 159
  18-months - smoking cigarettes: 'Several times' or 'a lot' | 33 | 22 | 28 | 18
  18-months - smoking cigarettes: 'None', 'once', or 'a few times' | 124 | 129 | 132 | 141
  18-months - using other drugs: number analyzed (Participants) | 157 | 151 | 160 | 159
  18-months - using other drugs: 'Several times' or 'a lot' | 28 | 23 | 26 | 19
  18-months - using other drugs: 'None', 'once', or 'a few times' | 129 | 128 | 134 | 140
Statistical Analysis 1: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; A sample size of 400 parents and children was calculated to yield 80% power to detect one or more differences between the intervention and control arms, of 45% in talking about alcohol, 20% about marijuana, and 20% about other drugs, using a two-sided Bonferroni-corrected 1.5% level of significance (based on estimates from the pilot trial); Test type: Superiority; p < 0.001, Generalized estimation — At 3 months: Parent-reported frequency of conversations on drinking alcohol; Prevalence Ratio (PR) = 2.86, 95% CI 2-sided [2.02 to 4.04]
Statistical Analysis 2: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p < 0.001, Generalized estimation — At 3 months: Parent-reported frequency of conversations on using e-cigarettes or vaping; Prevalence Ratio [PR] = 2.4, 95% CI 2-sided [1.67 to 3.45]
Statistical Analysis 3: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p < 0.001, Generalized estimation — At 3 months: Parent-reported frequency of conversations on using marijuana; Prevalence Ratio [PR] = 2.36, 95% CI 2-sided [1.62 to 3.43]
Statistical Analysis 4: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p < 0.001, Generalized estimation — At 3 months: Parent-reported frequency of conversations on smoking cigarettes; Prevalence Ratio [PR] = 3.45, 95% CI 2-sided [2.34 to 5.08]
Statistical Analysis 5: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p < 0.001, Generalized estimation — At 3 months: Parent-reported frequency of conversations on using other drugs; Prevalence Ratio [PR] = 2.47, 95% CI 2-sided [1.58 to 3.86]
Statistical Analysis 6: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p = 0.04, Generalized estimation — At 18 months: Parent-reported frequency of conversations on drinking alcohol; Prevalence Ratio [PR] = 1.45, 95% CI 2-sided [1.02 to 2.06]

2. Primary Outcome: Targeted Parent-child Communication on Substance Use
Description: An adapted version of the Targeted Parent-Child Communication about Alcohol Scale (Miller-Day et al, 2010) was used to assess targeted communication about alcohol and other drugs use. The ten-item assesses parents' agreement on having communication about substance use related topics and applying strategies parents may have discussed with their child. Items were assessed on a six-point Likert scale from "Strongly agree" to "Strongly disagree". Responses were dichotomized as "Agree" or "Strongly Agree" versus "Strongly Disagree" to "Somewhat Agree".
  This measure was reported by parents and children.
Time Frame: 3 months (short-term) and 18 months (long-term)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Substance Use Prevention Intervention | Substance Use Prevention Intervention - Children | Nutrition, Physical Activity, and Weight Talk Comparison | Nutrition, Physical Activity, and Weight Talk Comparison - Children
Number analyzed (Participants) | 181 | 181 | 185 | 185
Participants
  3 months - warned about the dangers: Agree | 162 | 147 | 126 | 143
  3 months - warned about the dangers: Disagree | 19 | 34 | 59 | 42
  3 months - talked about how to handle offers: Agree | 137 | 125 | 81 | 106
  3 months - talked about how to handle offers: Disagree | 44 | 56 | 104 | 79
  3 months - given rules to obey: Agree | 139 | 111 | 61 | 104
  3 months - given rules to obey: Disagree | 42 | 70 | 124 | 81
  3 months - not directly talked but given hints on not to use: Agree | 18 | 39 | 29 | 59
  3 months - not directly talked but given hints on not to use: Disagree | 163 | 142 | 156 | 126
  3 months - lectured or given speech: Agree | 71 | 83 | 41 | 68
  3 months - lectured or given speech: Disagree | 110 | 98 | 144 | 117
  3 months - made a comment if a character on TV is drinking/drunk: Agree | 83 | 84 | 57 | 64
  3 months - made a comment if a character on TV is drinking/drunk: Disagree | 98 | 97 | 128 | 121
  3 months - told stories of people who drink or have been drunk or use drugs: Agree | 112 | 60 | 86 | 60
  3 months - told stories of people who drink or have been drunk or use drugs: Disagree | 69 | 121 | 99 | 125
  3 months - told they would be disappointed: Agree | 88 | 77 | 47 | 71
  3 months - told they would be disappointed: Disagree | 93 | 104 | 138 | 114
  3 months - shown information about the dangers: Agree | 71 | 50 | 48 | 44
  3 months - shown information about the dangers: Disagree | 110 | 131 | 137 | 141
  3 months - asked about their thoughts or opinions: Agree | 144 | 101 | 83 | 81
  3 months - asked about their thoughts or opinions: Disagree | 37 | 80 | 102 | 104
  18 months - warned about the dangers: number analyzed (Participants) | 157 | 151 | 160 | 159
  18 months - warned about the dangers: Agree | 114 | 108 | 105 | 108
  18 months - warned about the dangers: Disagree | 43 | 43 | 55 | 51
  18 months - talked about how to handle offers: number analyzed (Participants) | 157 | 151 | 160 | 159
  18 months - talked about how to handle offers: Agree | 95 | 93 | 76 | 81
  18 months - talked about how to handle offers: Disagree | 62 | 58 | 84 | 78
  18 months - given rules to obey: number analyzed (Participants) | 157 | 151 | 160 | 159
  18 months - given rules to obey: Agree | 87 | 92 | 63 | 74
  18 months - given rules to obey: Disagree | 70 | 59 | 97 | 85
  18 months - not directly talked but given hints on not to use: number analyzed (Participants) | 157 | 151 | 160 | 159
  18 months - not directly talked but given hints on not to use: Agree | 18 | 22 | 27 | 49
  18 months - not directly talked but given hints on not to use: Disagree | 139 | 129 | 133 | 110
  18 months - lectured or given speech: number analyzed (Participants) | 157 | 151 | 160 | 159
  18 months - lectured or given speech: Agree | 50 | 62 | 32 | 47
  18 months - lectured or given speech: Disagree | 107 | 89 | 128 | 112
  18 months - made a comment if a character on TV is drinking/drunk: number analyzed (Participants) | 157 | 151 | 160 | 159
  18 months - made a comment if a character on TV is drinking/drunk: Agree | 69 | 47 | 50 | 52
  18 months - made a comment if a character on TV is drinking/drunk: Disagree | 88 | 104 | 110 | 107
  18 months - told stories of people who drink or have been drunk or use drugs: number analyzed (Participants) | 157 | 151 | 160 | 159
  18 months - told stories of people who drink or have been drunk or use drugs: Agree | 90 | 55 | 76 | 52
  18 months - told stories of people who drink or have been drunk or use drugs: Disagree | 67 | 96 | 84 | 107
  18 months - told they would be disappointed: number analyzed (Participants) | 157 | 151 | 160 | 159
  18 months - told they would be disappointed: Agree | 56 | 59 | 41 | 52
  18 months - told they would be disappointed: Disagree | 101 | 92 | 119 | 107
  18 months - shown information about the dangers: number analyzed (Participants) | 157 | 151 | 160 | 159
  18 months - shown information about the dangers: Agree | 56 | 36 | 38 | 37
  18 months - shown information about the dangers: Disagree | 101 | 115 | 122 | 122
  18 months - asked about their thoughts or opinions: number analyzed (Participants) | 157 | 151 | 160 | 159
  18 months - asked about their thoughts or opinions: Agree | 99 | 64 | 84 | 57
  18 months - asked about their thoughts or opinions: Disagree | 58 | 87 | 76 | 102
Statistical Analysis 1: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p < 0.001, Generalized estimation — At 3 months: Parent-reported "have warned your child about the dangers of drinking alcohol and using drugs"; Prevalence Ratio (PR) = 1.31, 95% CI 2-sided [1.18 to 1.45]
Statistical Analysis 2: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p < 0.001, Generalized estimation — At 3 months: Parent-reported 'have talked to your child about how to handle offers of alcoholic drinks and drugs'; Prevalence Ratio [PR] = 1.55, 95% CI 2-sided [1.32 to 1.83]
Statistical Analysis 3: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p < 0.001, Generalized estimation — At 3 months: Parent-reported 'have given your child rules to obey about drinking alcohol and using drugs'; Prevalence Ratio [PR] = 2.13, 95% CI 2-sided [1.73 to 2.63]
Statistical Analysis 4: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p = 0.001, Generalized estimation — At 3 months: Parent-reported 'have lectured or given your child a speech about drinking alcohol and using drugs'; Prevalence Ratio [PR] = 1.67, 95% CI 2-sided [1.25 to 2.25]
Statistical Analysis 5: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p < 0.001, Generalized estimation — At 3 months: Parent-reported 'have made a comment to your child about how drinking alcohol and using drugs is bad if a character on TV is drinking or drunk'; Prevalence Ratio [PR] = 1.51, 95% CI 2-sided [1.21 to 1.90]
Statistical Analysis 6: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p = 0.008, Generalized estimation — At 3 months: Parent-reported 'have told your child stories of people who drink alcohol, have been drunk, or use drugs'; Prevalence Ratio [PR] = 1.25, 95% CI 2-sided [1.06 to 1.47]
Statistical Analysis 7: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p < 0.001, Generalized estimation — At 3 months: Parent-reported 'have told your child you would be disappointed in her/him if they were to drink alcohol or use drugs'; Prevalence Ratio [PR] = 1.65, 95% CI 2-sided [1.29 to 2.10]
Statistical Analysis 8: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p < 0.001, Generalized estimation — At 3 months: Parent-reported 'have shown your child information on the web, TV, or in the news about the dangers of drinking alcohol and using drugs'; Prevalence Ratio [PR] = 1.64, 95% CI 2-sided [1.24 to 2.15]
Statistical Analysis 9: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p < 0.001, Generalized estimation — At 3 months: Parent-reported 'have asked your child about their thoughts and opinions about drinking alcohol and using drugs'; Prevalence Ratio [PR] = 1.65, 95% CI 2-sided [1.40 to 1.93]
Statistical Analysis 10: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p = 0.003, Generalized estimation — At 18 months: Parent-reported 'have given your child rules to obey about drinking alcohol and using drugs'; Prevalence Ratio [PR] = 1.40, 95% CI 2-sided [1.12 to 1.74]
Statistical Analysis 11: Comparison: Substance Use Prevention Intervention vs Nutrition, Physical Activity, and Weight Talk Comparison; Test type: Superiority; p = 0.01, Generalized estimation — At 18 months: Parent-reported 'have made a comment to your child about how drinking alcohol and using drugs is bad if a character on TV is drinking or drunk'; Prevalence Ratio [PR] = 1.38, 95% CI 2-sided [1.06 to 1.78]

3. Primary Outcome: Parent-child Audio-recorded Conversations About Substance Use
Description: The prompts, modeled after the Family Assessment Task (FAsTask) where parents and adolescents have a conversation about substance use and related behaviors, were developed by the study team (Spirito et al, 2011). The same prompts are used at each time point. The sub-scales (expectations, messaging, communication style, and strategies) range from 1 to 9 (higher values represent a higher quality conversation compared to lower values). The overall combined score ranges from 4 to 36 (higher values represent a higher quality conversation compared to lower values).
Time Frame: 12 months
Population: Sample sizes differ at each follow-up based on how many parents and children completed the audio submission.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Substance Use Prevention Intervention | Nutrition, Physical Activity, and Weight Talk Comparison
Number analyzed (Participants) | 90 | 86
score
  Expectations | 3.5 (2.1) | 3.2 (1.9)
  Messaging | 4.7 (1.3) | 4.6 (1.3)
  Communication style | 5.5 (1.6) | 5.5 (1.5)
  Strategies | 2.4 (1.8) | 2.2 (1.5)
  Overall combined score | 16 (4.0) | 15.5 (3.5)

4. Primary Outcome: Quality of Video-recorded Family Mealtime Interactions
Description: The mean quality of mealtime interactions is measured using various scales from the Iowa Family Interaction Rating Scales (IFIRS) coding system: Dyadic Interaction Scales, Dyadic Relationship Scales, Group Interactions Scales, and Parenting Scales. Observed behaviors from 3 video-recorded family meals are assessed and scored on a 9-point scale. A higher score indicates coders observed a higher intensity and/or frequency of the construct in the video-recorded family meals. Each IFIRS scale is scored individually, and the average across the 3 family meals is reported. The items were organized into four subscales: Communication (range: 4-36), Parenting Style (range: 5-45), Dyad Relationship (range: 5-45), and Group Enjoyment (range: 1-9).
Time Frame: 12 months
Population: Sample sizes differ at each follow-up based on how many parents and children completed the video submission.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Substance Use Prevention Intervention | Nutrition, Physical Activity, and Weight Talk Comparison
Number analyzed (Participants) | 90 | 92
score
  Parent communication | 28.9 (0.3) | 28.6 (0.3)
  Parenting style | 30.3 (0.2) | 30.1 (0.2)
  Dyad relationship | 25.7 (0.3) | 25.8 (0.3)
  Group enjoyment | 4.5 (0.1) | 4.2 (0.1)

5. Primary Outcome: Child Substance Use Expectancies (Alcohol)
Description: Positive and negative expectancies about the affective, cognitive, and behavioral effects of alcohol use will be assessed with the Alcohol Expectancy Questionnaire-Adolescent Form, short version. The tool is comprised of 27 items, each with response options ranging from (1) Strongly Disagree to (6) Strongly Agree. Questions 6, 9, 17, and 26 are scored in opposite direction before they are included in the negative sub-scale (remaining items are included in the positive sub-scale). Sub-scales are created by averaging the items and range from 1 to 6. A higher score on the positive expectancies scale indicates a greater belief that alcohol has desirable effects, and a higher score on the negative expectancies scale indicates a greater belief that alcohol has undesirable effects.
  This measure was reported by children only.
Time Frame: 18 months
Population: Sample sizes differ based on how many children completed the survey at each follow-up.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Substance Use Prevention Intervention - Children | Nutrition, Physical Activity, and Weight Talk Comparison - Children
Number analyzed (Participants) | 129 | 140
score
  Positive expectancies | 2.55 (0.08) | 2.53 (0.07)
  Negative expectancies | 4.24 (0.09) | 4.23 (0.09)

6. Primary Outcome: Child Substance Use Expectancies (Cigarettes)
Description: Positive and negative expectancies about the affective, cognitive, and behavioral effects of cigarette use will be assessed with the Positive and Negative Outcome Expectancies of Smoking scale. The tool comprises 12 items, each with response options ranging from (1) Strongly Disagree to (6) Strongly Agree. The tool has two subscales (positive expectancies, determined by 7 questions; negative expectancies, determined by 5 questions). Summary scores for both the positive and negative expectancies are created. Summary score values range from 0-7 for positive, 0-5 for negative expectancies. Higher score on positive expectancies scale indicates a greater belief that there are positive outcomes of smoking. Higher score on negative expectancies scale indicates a greater belief in negative consequences of smoking.
  This measure was reported by children only.
Time Frame: 18 months
Population: Sample sizes differ based on how many children completed the survey at each follow-up.
Measure: Mean (Standard Error); unit: score
Groups:
- Substance Use Prevention Intervention - Children: Parents were given a handbook specific to the gender of their child that provides information and advice communication and substance use prevention. Parents then participated in a one-hour session with an interventionist where the main points in the handbook were reviewed and they filled out an action plan on how to make changes in communication about substances with their child. The interventionist also provided parents with a referral packet. Two weeks after the live session, participants had a half-hour follow-up phone call with the same study interventionist. For the home-based component, parents received two messages each week with reminders and tips that reinforce the information covered in the handbook. Finally, participants received a magnet about the importance of family meals that they were instructed to put on their refrigerators.
- Nutrition, Physical Activity, and Weight Talk Comparison - Children: For the comparison condition, after the baseline assessment, parents received a handbook on nutrition and physical activity entitled: "Healthy Eating & Physical Activity Across Your Lifespan: Helping your Child - Tips for Parents". This handbook, which is adapted from the handbook developed by the National Institute of Diabetes and Digestive and Kidney Diseases and the Weight Control Information Network, is approximately the same length as the intervention handbook and is available in English and Spanish. It is given with an insert on reducing weight talk and weight teasing in the family. Parents also received a magnet with a message about nutrition and exercise. To control for contact time, these participants met live with a study staff member two weeks after receiving the handbook, completed an action plan, and had the 30-minute call, as well as receive two text messages twice per week for 13 weeks with tips and reminders from the comparison handbook and insert.
Arm/Group | Substance Use Prevention Intervention - Children | Nutrition, Physical Activity, and Weight Talk Comparison - Children
Number analyzed (Participants) | 133 | 143
score
  Positive expectancies | 1.68 (0.05) | 1.57 (0.05)
  Negative expectancies | 5.15 (0.07) | 5.22 (0.07)

7. Primary Outcome: Child Substance Use Expectancies (Marijuana)
Description: Positive and negative expectancies about the affective, cognitive, and behavioral effects of marijuana use will be assessed with an adapted version of the Marijuana Effect Expectancies Questionnaire - Brief. The tool comprises three standalone subscales (Relaxation/Tension Reduction, Cognitive/Behavioral Impairment, Global Negative Effects) for a total of 27 items. Each item has responses ranging from (1) Strongly Disagree to (6) Strongly Agree. Scores for each subscale are calculated by averaging item scores within that subscale. Each subscale score range is from 1 - 6. Higher scores on each scale indicate greater expectations positive expectancies (Relaxation/Tension Reduction) and negative expectancies (Cognitive/Behavioral Impairment and Global Negative Effects) associated with marijuana use.
  This measure was reported by children only.
Time Frame: 18 months
Population: Sample sizes differ based on how many children completed the survey at each follow-up.
Measure: Mean (Standard Error); unit: score
Arm/Group | Substance Use Prevention Intervention - Children | Nutrition, Physical Activity, and Weight Talk Comparison - Children
Number analyzed (Participants) | 128 | 140
score
  Positive expectancies | 2.69 (0.1) | 2.73 (0.1)
  Negative expectancies | 4.04 (0.12) | 4.16 (0.12)

8. Primary Outcome: Child Affiliation With Substance-using Peers
Description: Using an item from the Monitoring the Future study, children will be asked how many of their friends they think use substances. The item is repeated for each substance.
  This measure was reported by children only.
Time Frame: 18 months
Population: Sample sizes differ based on how many children completed the survey at each follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Substance Use Prevention Intervention - Children | Nutrition, Physical Activity, and Weight Talk Comparison - Children
Number analyzed (Participants) | 148 | 148
Participants
  How many of your friends do you estimate occassionally drink alcohol?: number analyzed (Participants) | 145 | 141
  How many of your friends do you estimate occassionally drink alcohol?: Some to most | 21 | 15
  How many of your friends do you estimate occassionally drink alcohol?: None | 124 | 126
  How many of your friends do you think smoke cigarettes?: number analyzed (Participants) | 148 | 147
  How many of your friends do you think smoke cigarettes?: Some to most | 11 | 4
  How many of your friends do you think smoke cigarettes?: None | 137 | 143
  How many of your friends do you think use marijuana?: number analyzed (Participants) | 146 | 148
  How many of your friends do you think use marijuana?: Some to most | 15 | 11
  How many of your friends do you think use marijuana?: None | 131 | 137
  How many of your friends do you estimate occassionally use e-cigarettes or vapes?: number analyzed (Participants) | 146 | 142
  How many of your friends do you estimate occassionally use e-cigarettes or vapes?: Some to most | 29 | 23
  How many of your friends do you estimate occassionally use e-cigarettes or vapes?: None | 117 | 119
  How many of your friends do you think use other drugs?: number analyzed (Participants) | 144 | 141
  How many of your friends do you think use other drugs?: Some to most | 4 | 2
  How many of your friends do you think use other drugs?: None | 140 | 139

9. Primary Outcome: Child Willingness to Use Substances
Description: Child willingness to use substances will be assessed through three items adapted from the measure combining intention and willingness originally developed for tobacco and amphetamines found in Gibbons et al. (1998) Reasoned Action and Social Reaction: Willingness and Intention as Independent Predictors of Health Risk. The three items will be asked for each substance. Each item has response options ranging from (1) Not at all likely to (6) Very likely. Response options are transformed to binary format such that 0 represents (1) Not at all likely and 1 represents (2) Unlikely to (6) Very Likely. The three binary items are then averaged for each substance and scores range from 0 to 1 (0 being not willing at all and 1 being somewhat to very likely willing to use the substance).
  This measure was reported by children only.
Time Frame: 18 months
Population: Sample sizes differ based on how many children completed the survey at each follow-up.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Substance Use Prevention Intervention - Children | Nutrition, Physical Activity, and Weight Talk Comparison - Children
Number analyzed (Participants) | 149 | 156
score
  Alcohol - Willingness to use: number analyzed (Participants) | 149 | 154
  Alcohol - Willingness to use | 0.27 (0.64) | 0.26 (0.63)
  Cigarettes - Willingness to use: number analyzed (Participants) | 148 | 156
  Cigarettes - Willingness to use | 0.22 (0.61) | 0.13 (0.41)
  Cannabis - Willingness to use: number analyzed (Participants) | 149 | 154
  Cannabis - Willingness to use | 0.24 (0.66) | 0.15 (0.45)
  E-cigarettes or vaping - Willingness to use: number analyzed (Participants) | 148 | 153
  E-cigarettes or vaping - Willingness to use | 0.34 (0.85) | 0.21 (0.56)
  Other drugs - Willingness to use: number analyzed (Participants) | 138 | 144
  Other drugs - Willingness to use | 0.12 (0.44) | 0.17 (0.49)

10. Primary Outcome: Child Intentions to Use Substances
Description: One item from the Youth Alcohol and Drug Survey will assess child's intention to use substances in the next 30 days. The question is asked for each substance and has the response options 'No', 'Probably No', 'Probably Yes', 'Yes'. Response options are dichotomized to (1) No [which includes 'No' and 'Probably No'] and (2) Yes [which includes 'Probably Yes' and 'Yes'].
  This measure was reported by children only.
Time Frame: 18 months
Population: Sample sizes differ based on how many children completed the survey at each follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Substance Use Prevention Intervention - Children | Nutrition, Physical Activity, and Weight Talk Comparison - Children
Number analyzed (Participants) | 147 | 148
Participants
  Alcohol - Plan to use in the next 30 days: number analyzed (Participants) | 147 | 146
  Alcohol - Plan to use in the next 30 days: Yes | 0 | 0
  Alcohol - Plan to use in the next 30 days: No | 147 | 146
  Cigarettes - Plan to use in the next 30 days: Yes | 0 | 0
  Cigarettes - Plan to use in the next 30 days: No | 147 | 148
  Cannabis - Plan to use in the next 30 days: number analyzed (Participants) | 147 | 147
  Cannabis - Plan to use in the next 30 days: Yes | 0 | 0
  Cannabis - Plan to use in the next 30 days: No | 147 | 147
  E-cigarettes or vapes - Plan to use in the next 30 days: Yes | 1 | 1
  E-cigarettes or vapes - Plan to use in the next 30 days: No | 146 | 147
  Other drugs - Plan to use in the next 30 days: number analyzed (Participants) | 144 | 140
  Other drugs - Plan to use in the next 30 days: Yes | 0 | 0
  Other drugs - Plan to use in the next 30 days: No | 144 | 140

11. Secondary Outcome: Pre/Early-adolescent Substance Use Initiation
Description: Substance use initiation for each substance will be assessed with three items from the Drug Use Questionnaire. The items will be asked for each substance. Child responds Yes/No to the "have you ever used [substance]?" question.
  This measure was reported by children only.
Time Frame: 18 months
Population: Sample sizes differ based on how many children completed the survey at each follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Substance Use Prevention Intervention - Children | Nutrition, Physical Activity, and Weight Talk Comparison - Children
Number analyzed (Participants) | 187 | 182
Participants
  Alcohol: Yes | 14 | 9
  Alcohol: No | 173 | 173
  Cigarettes: Yes | 3 | 2
  Cigarettes: No | 184 | 180
  Cannabis: Yes | 9 | 3
  Cannabis: No | 178 | 179
  E-cigarettes or vaping: Yes | 13 | 6
  E-cigarettes or vaping: No | 174 | 176
  Other drugs: Yes | 1 | 1
  Other drugs: No | 186 | 181

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 24 months (from randomization through study completion date) for parent and child participants, and no adverse events were reported.
Groups:
- Substance Use Prevention Intervention - Parents: Parents were given a handbook specific to the gender of their child that provides information and advice communication and substance use prevention. Parents then participated in a one-hour session with an interventionist where the main points in the handbook were reviewed and they filled out an action plan on how to make changes in communication about substances with their child. The interventionist also provided parents with a referral packet. Two weeks after the live session, participants had a half-hour follow-up phone call with the same study interventionist. For the home-based component, parents received two messages each week with reminders and tips that reinforce the information covered in the handbook. Finally, participants received a magnet about the importance of family meals that they were instructed to put on their refrigerators.
  The SUPPER Project: Substance Use Promoted by Eating family meals Regularly
- Nutrition, Physical Activity, and Weight Talk Comparison - Parents: For the comparison condition, after the baseline assessment, parents received a handbook on nutrition and physical activity entitled: "Healthy Eating & Physical Activity Across Your Lifespan: Helping your Child - Tips for Parents". This handbook, which is adapted from the handbook developed by the National Institute of Diabetes and Digestive and Kidney Diseases and the Weight Control Information Network, is approximately the same length as the intervention handbook and is available in English and Spanish. It is given with an insert on reducing weight talk and weight teasing in the family. Parents also received a magnet with a message about nutrition and exercise. To control for contact time, these participants met live with a study staff member two weeks after receiving the handbook, completed an action plan, and had the 30-minute call, as well as receive two text messages twice per week for 13 weeks with tips and reminders from the comparison handbook and insert.
  Improving nutrition and physical activity among youth: A brief intervention focused on improving nutrition and physical activity among youth
Arm/Group | Substance Use Prevention Intervention - Parents | Substance Use Prevention Intervention - Children | Nutrition, Physical Activity, and Weight Talk Comparison - Parents | Nutrition, Physical Activity, and Weight Talk Comparison - Children
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/201 | 0/201 | 0/201
Serious Adverse Events (participants affected / at risk) | 0/201 | 0/201 | 0/201 | 0/201
Other Adverse Events (participants affected / at risk) | 0/201 | 0/201 | 0/201 | 0/201

LIMITATIONS AND CAVEATS:
It was hypothesized a priori that the intervention's effects would not be able to be determined through differences in child-reported substance use outcomes, since the prevalence of substance use in this age group is historically very low.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-11-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT03925220/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT03925220/SAP_001.pdf
  • Informed Consent Form (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT03925220/ICF_002.pdf